CLINICAL TRIAL: NCT03396484
Title: Methyldopa for Reduction of DQ8 Antigen Presentation in At-Risk Subjects for Type 1 Diabetes Mellitus
Brief Title: Methyldopa for Reduction of DQ8 Antigen Presentation in At-Risk Subjects for Type 1 Diabetes
Acronym: TN-23
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not begun due to continued laboratory work on the feasibility of outcome measures.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Methyldopa; UC4DK106993 (NIH); UC4DK117009 (NIH)
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Type1 Diabetes Mellitus
Keywords: TrialNet
MeSH Terms: interventions — Methyldopa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methyldopa (Experimental): Adults: methyldopa 500mg twice daily for one week and then increased to 500mg three times a day
  Children: methyldopa dose based on weight twice daily for one week then increased to three times a day
  Interventions: Drug: Methyldopa
- Placebo (Placebo Comparator): Inactive agent to match active drug in appearance and dose frequency.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methyldopa — Tablet for oral dosing
  Other Names: Aldomet
  Arms: Methyldopa
Drug: Placebo — Tablet for oral dosing
  Arms: Placebo

SUMMARY:
A study is to see if methyldopa can change the immune system's attack on insulin producing cells in people at early stages of type 1 diabetes.

DETAILED DESCRIPTION:
The study is a randomized, double blinded, placebo-controlled, multi-center crossover clinical trial.

Eligible subjects will be randomized in a 1:1 allocation ratio to one of two treatment schedules: first methyldopa then placebo vs. first placebo then methyldopa.

The study objective is to assess the safety, efficacy, and mode of action of methyldopa to reduce DQ8 antigen presentation in individuals at Stage 1 and 2 of type 1 diabetes (T1D).

ELIGIBILITY:
Inclusion Criteria:

* Participant in TrialNet Pathway to Prevention Study (TN01)
* Willing to provide Informed Consent or, if the subject is <18 years of age, have a parent or legal guardian provide Informed Consent
* Confirmed positive for one or more autoantibodies, one of which is insulin autoantibody (mIAA)
* Positive for at least one gene encoding HLA-DQ8 (DQB*0302)
* If a female participant with reproductive potential, willing to avoid pregnancy and undergo pregnancy testing prior to randomization and during the study
* Have normal or abnormal glucose tolerance on OGTT performed within 7 weeks of randomization

Exclusion Criteria:

* Inability or unwillingness of a participant to give written informed consent or comply with study protocol
* History of clinically significant anemia or Hemoglobin <10 g/dl
* Evidence of liver dysfunction
* History of renal insufficiency
* History of symptomatic hypotension including positional hypotension
* Systolic BP < 100 mmHg for adults or blood pressure < 5th percentile for age/height/gender in children and adolescents
* Use of a treatment that is known to cause a significant, ongoing change in the course of diabetes or immunologic status, within 4 weeks prior to participation. This includes high-dose inhaled, extensive topical or systemic glucocorticoids
* Females who are pregnant at the time of screening, breastfeeding or unwilling to defer pregnancy during the 16-month study period. (Female participant must be at least 100 days postpartum before enrollment into study)
* Unable to avoid concurrent antihypertensive medications, monoamine oxidase (MAO) inhibitors, lithium, or medications containing ferrous sulfate or ferrous gluconate
* Unable to avoid medications that affect stomach pH, such as proton pump inhibitors or histamine H2 receptor blockers
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
DQ8 Antigen Presentation | 6 months after initiation of treatment
  insulin peptide-specific DQ8 antigen presentation

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet

REFERENCES:
- See also: TrialNet Public Website — https://www.trialnet.org/